CLINICAL TRIAL: NCT02411994
Title: Pyronaridine-artesunate and Artemether-lumefantrine for the Treatment of Paediatric Uncomplicated Falciparum Malaria in Western Kenya
Brief Title: Pyronaridine-artesunate and Artemether-lumefantrine for the Treatment of Paediatric Malaria
Acronym: PAAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royal Tropical Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KIT601714
Record Dates: First submitted 2015-04-03; First posted 2015-04-08 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pyronaridine-artesunate (Experimental): pyronaridine-artesunate: recommended dose according to body weight, once a day for three days.
  Interventions: Drug: Pyronaridine-artesunate
- Artemether-lumefantrine (Active Comparator): artemether-lumefantrine: recommended dose according to body weight, twice a day for three days.
  Interventions: Drug: Artemether-lumefantrine combination

INTERVENTIONS:
Drug: Pyronaridine-artesunate
  Other Names: Pyramax
  Arms: Pyronaridine-artesunate
Drug: Artemether-lumefantrine combination
  Other Names: Coartem
  Arms: Artemether-lumefantrine

SUMMARY:
The purpose of this study is to determine the efficacy of pyronaridine-artesunate and artemether-lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria in Kenyan children.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 months and 12 years old, with a body weight of ≥5 kg;
* Living in the catchment area of the study (within a radius of ~10 km from St. Jude's Clinic, Mbita, Kenya);
* Having microscopically confirmed P. falciparum mono-infection (asexual parasite density 1,000-200,000 µL-1).

Exclusion Criteria:

* Signs and symptoms of severe malaria (according to WHO criteria for severe malaria, (WHO 2012)) or any other severe illness necessitating parenteral treatment;
* Mixed Plasmodium infection;
* Clinically suspected (oedema, jaundice and/or ascites) or reported hepatic and/or renal impairment (any cause, as reported by parents/guardians and/or evident from medical history);
* Having anaemia with an Hb <6 g/dL;
* Evidence of severe malnutrition (severe wasting: z-score weight for age <-3 and severe stunting: z-score height for age <-3 (WHO 2009b));
* Having received anti-malarial therapy in the previous two weeks;
* Known history of hypersensitivity, allergic or adverse reactions to artesunate, artemether-lumefantrine or other artemisinins;
* Participating in other anti-malarial drug intervention studies;
* Previous participation in the PAAL study, e.g. in the previous transmission season (each individual child can only take part in this study once);
* Not being available for follow-up.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 197 (Actual)
Dates: Start 2015-10; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
PCR-corrected adequate clinical and parasitological response (ACPR) | day 28 after initial dose

SECONDARY OUTCOMES:
PCR-corrected adequate clinical and parasitological response (ACPR) | day 42 after initial dose
crude adequate clinical and parasitological response (ACPR) | day 28, day 42 after initial dose
parasite clearance time | up to 7 days after initial dose
gametocyte clearance time | up to 7 days after initial dose
transmission potential to mosquitos | day 7 after initial dose

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Sawa, MD, PhD, Principal Investigator — International Centre of Insect Physiology and Ecology (ICIPE)
Locations (1):
- St. Jude's Clinic, ICIPE, Mbita, Kenya

REFERENCES:
- [Derived] Roth JM, Sawa P, Omweri G, Osoti V, Makio N, Bradley J, Bousema T, Schallig HDFH, Mens PF. Plasmodium falciparum gametocyte dynamics after pyronaridine-artesunate or artemether-lumefantrine treatment. Malar J. 2018 Jun 4;17(1):223. doi: 10.1186/s12936-018-2373-7. PMID 29866116
- [Derived] Roth JM, Sawa P, Makio N, Omweri G, Osoti V, Okach S, Choy F, Schallig HDFH, Mens P. Pyronaridine-artesunate and artemether-lumefantrine for the treatment of uncomplicated Plasmodium falciparum malaria in Kenyan children: a randomized controlled non-inferiority trial. Malar J. 2018 May 15;17(1):199. doi: 10.1186/s12936-018-2340-3. PMID 29764419